#### Official Title:

Efficacy of Propofol Combination with either Ketamine, Dexmedetomidine or Midazolam for Sedation during Upper Gastrointestinal Endoscopic Procedures: A Prospective, Randomized, Comparative Study

#### **NCT Number:**

Pending (to be assigned by ClinicalTrials.gov)

## **Document Type:**

Statistical analysis plan

### Version/Date:

Version 1.0 – July 29, 2024



# Methodological Approach of a Research Protocol A Review Checklist

<u>Title of the Research:</u> Efficacy of Propofol Combination with either Ketamine, Dexmedetomidine or Midazolam for Sedation during Upper Gastrointestinal Endoscopic Procedures: A Prospective, Randomized, Comparative Study

Name of Researcher: Hazem Mohamed Sabry Abdelaziz

Specialty: Anesthesia

Type of Research: MD degree

#### I- Research Objective

a. Well formulated objective:  $\sqrt{\phantom{a}}$ 

**Proposed reformulated objective:** To compare the following sedative combinations (ketamine-propofol, dexmedetomidine-propofol and midazolam-propofol) as regard the recovery time for patients undergoing elective upper gastrointestinal endoscopic procedures.

Objective conforming with study design  $\sqrt{\phantom{a}}$ 

· II-Study Design Review

- a. Type of Study Design: ----
- b. Proposed study design: Three Arms Randomized Clinical Trial

#### III- Sample Size:

Using G power software for sample size calculation: setting power at 80% and  $\alpha$  error at 5%, it is estimated that a sample size of 66 patients undergoing elective upper gastrointestinal endoscopic procedures (22 patients receiving ketamine-propofol, 22 patients receiving dexmedetomidine-propofol, and 22 patients receiving midazolam-propofol combinations) will be needed to detect a statistically significant difference between the three groups as regards the recovery time in minutes, assuming a large effect size (f=0.40) regarding *Tekeli et al.*, 2020, using F test (ANOVA: fixed effects, omnibus, one-way).

Assuming that the dropout is of 10%, a sample size of at least 75 patients undergoing elective upper gastrointestinal endoscopic procedures (25

patients per group) will be needed.

IV- Missed Items to be added: -

Name of Reviewer: Dr. Shaimaa Samy Yousef

of Medicine Ain Shows University

Presented for Medical Research Ethical Committee at Faculty of Medicine Ain Shams University

Review Checklist